CLINICAL TRIAL: NCT02446132
Title: A Phase 3, Multicenter, Long Term, Extension Study of the Safety and Efficacy of AVP-786 (Deuterated [d6] Dextromethorphan Hydrobromide [d6-DM]/Quinidine Sulfate [Q]) for the Treatment of Agitation in Patients With Dementia of the Alzheimer's Type
Brief Title: Long Term, Extension Study of the Safety and Efficacy of AVP-786 for the Treatment of Agitation in Patients With Dementia of the Alzheimer's Type
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The AVP-786 program was discontinued, the recruitment was stopped and all participants are no longer being examined or receiving intervention.
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-AVP-786-303; 2017-002455-29 (EudraCT Number)
Record Dates: First submitted 2015-05-11; First posted 2015-05-18 (Estimated); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-08

CONDITIONS: Agitation in Patients With Dementia of the Alzheimer's Type

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AVP-786 18 milligrams (mg) (Experimental): Participants who received AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) capsules in the previous studies 15-AVP-786-301 (NCT02442765), 15-AVP-786-302 (NCT02442778), or 17-AVP-786-305 (NCT03393520) continued to receive AVP-786-18 (d6-DM 18 mg/Q 4.9 mg), capsules, twice a day for 52 weeks in the current study.
  Interventions: Drug: AVP-786
- AVP-786 28 mg (Experimental): Participants who received AVP-786-28 (d6-DM 28 mg/Q 4.9 mg) capsules in the previous studies 15-AVP-786-301 (NCT02442765), 15-AVP-786-302 (NCT02442778), or 17-AVP-786-305 (NCT03393520) continued to receive AVP-786-28 (d6-DM 28 mg/Q 4.9 mg), capsules, twice a day for 52 weeks in the current study.
  Interventions: Drug: AVP-786
- AVP-786 42.63 mg (Experimental): Participants who received placebo in the previous studies 15-AVP-786-301 (NCT02442765), 15-AVP-786-302 (NCT02442778), or 17-AVP-786-305 (NCT03393520) and those who had delayed enrolment, started AVP-786-28/4.9 (d6-DM 28 mg/Q 4.9 mg) in the current study and were eventually titrated to receive AVP-786-42.63/4.9 (d6-DM 42.63 mg/Q 4.9 mg) capsules, twice a day for 52 weeks.
  Interventions: Drug: AVP-786

INTERVENTIONS:
Drug: AVP-786

SUMMARY:
This was an extension study of the Phase 3 Studies 15-AVP-786-301, 15-AVP-786-302, and 17-AVP-786-305.

DETAILED DESCRIPTION:
Eligible participants for this study had successfully completed Studies 15-AVP-786-301, 15-AVP-786-302, 12-AVR-131, or 17-AVP-786-305.

Study medication was administered orally twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Participant has successfully completed Studies 15-AVP-786-301, 15-AVP-786-302, 12-AVR-131, or 17-AVP-786-305. (Note: A delay in enrollment may include delays associated with COVID-19 restrictions.)
* Participants with a diagnosis of probable Alzheimer's Disease (AD) according to the 2011 National Institute on Aging-Alzheimer's Association (NIA-AA) working group criteria
* Either out-patients or residents of an assisted-living facility or a skilled nursing home
* Participants who delay enrollment must have clinically significant, moderate/severe agitation at least 2 weeks prior to baseline
* Participants who delay enrollment must have a diagnosis of agitation that must meet the International Psychogeriatric Association (IPA) provisional definition of agitation
* Participants who delay enrollment must have a Clinical Global Impression of Severity of Illness (CGIS) score assessing Agitation of ≥ 4 (moderately ill) at screening and baseline
* Participants who delay enrollment must have a Mini-Mental State Examination (MMSE) score between 6 and 26 (inclusive) at screening and baseline

Exclusion Criteria:

* Participants with co-existent clinically significant or unstable systemic diseases that could confound the interpretation of the safety results of the study (e.g., malignancy, poorly controlled diabetes, poorly controlled hypertension, unstable pulmonary, renal or hepatic disease, unstable ischemic cardiac disease, dilated cardiomyopathy, or unstable valvular heart disease)
* Participants determined to have a high imminent risk of falls during the study based on a clinical evaluation by the investigator
* Participants who are currently using or were on NUEDEXTA® in the 2 weeks preceding baseline

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1197 (Actual)
Dates: Start 2015-11-13 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (227):
- United States (171):
  - MD First Research, LLC Site #767, Chandler, Arizona
  - NoesisPharma, LLC, Phoenix, Arizona
  - Perseverance Research Center, LLC, Scottsdale, Arizona
  - Health Initiatives Research, Fayetteville, Arkansas
  - Advanced Research Center, Inc. Site #835, Anaheim, California
  - ATP Clinical Research, Inc. Site #763, Costa Mesa, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Irvine Center for Clinical Research, Irvine, California
  - Sheenath Clinical Service Site #770, Lakewood, California
  - Torrance Clinical Research Institute, Inc. Site #826, Lomita, California
  - Collaborative Neuroscience Network, LLC., Long Beach, California
  - Alliance for Wellness, Inc dba Alliance for Research Site #789, Long Beach, California
  - NRC Research Institute, Orange, California
  - California Neurological Services, Panorama City, California
  - Havana Research Institute Site 787, Pasadena, California
  - Havana Research Institute, Pasadena, California
  - Pacific Research Network, Inc. #1, San Diego, California
  - Pacific Research Network, Inc. #2, San Diego, California
  - HB Clinical Trials Inc., Santa Ana, California
  - Syrentis Clinical Research, Santa Ana, California
  - Viking Clinical Research, Temecula, California
  - Lytle and Weiss, PLLC dba Clinical Trials of the Rockies, Denver, Colorado
  - Coastal Connecticut Research, LLC, New London, Connecticut
  - Research Center for Clinical Studies, Inc., Norwalk, Connecticut
  - Neurology of Central Florida Rsch Ctr Site #803, Altamonte Springs, Florida
  - JEM Research Institute, Atlantis, Florida
  - Negron Research Services / Humanity Clinical Research Site# 766, Aventura, Florida
  - SFM Clinical Research, LLC Site #563, Boca Raton, Florida
  - Bradenton Research Center Site #834, Bradenton, Florida
  - Clinical Research Of Brandon, LLC Site #838, Brandon, Florida
  - Clinical Research of Brandon, Brandon, Florida
  - Meridien Research, Brooksville, Florida
  - Quantum Laboratories, Inc., Deerfield Beach, Florida
  - Moonshine Research Center, Inc, Doral, Florida
  - Science Connections, LLC Site #814, Doral, Florida
  - Finlay Medical Research Corp, Greenacres City, Florida
  - Direct Helpers Research Center #801, Hialeah, Florida
  - Indago Research & Health Center, Inc., Hialeah, Florida
  - New Life Medical Research Center, Inc., Hialeah, Florida
  - Reliable Clinical Research,LLC, Hialeah, Florida
  - Research in Miami, Inc, Hialeah, Florida
  - The Research Center, Inc, Hialeah, Florida
  - Berma Research Group, Hialeah, Florida
  - Galiz Research, Hialeah, Florida
  - Maxblue Institute, Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Alphab Global Research #793, Jupiter, Florida
  - SIH Research, LLC, Kissimmee, Florida
  - Alzheimer's Research and Treatment Center #1, Lake Worth, Florida
  - Alzheimer's Research and Treatment Center #2, Lake Worth, Florida
  - Alzheimer's Research and Treatment Center #3, Lake Worth, Florida
  - Meridien Research Site #558, Lakeland, Florida
  - Innovative Clinical Research, Inc. Site #819, Lauderhill, Florida
  - Homestead Associates in Research Site# 797, Miami, Florida
  - Premier Clinical Research Institute, Inc. #1, Miami, Florida
  - Premier Clinical Research Institute, Inc. #2, Miami, Florida
  - Central Miami Medical Institute Site #798, Miami, Florida
  - Global Medical Institutes, LLC, Miami, Florida
  - Optimus U Corp, Miami, Florida
  - Project 4 Research #1, Miami, Florida
  - Project 4 Research #2, Miami, Florida
  - BioMed Research Institute, Miami, Florida
  - Finlay Medical Research Corp Site #552, Miami, Florida
  - First Class Medical Services Site #807, Miami, Florida
  - CCM Clinical Research Group, Miami, Florida
  - Innova Clinical Trials, Miami, Florida
  - Advance Medical Research Center #1, Miami, Florida
  - Advance Medical Research Center #2, Miami, Florida
  - Dade Research Center Llc, Miami, Florida
  - Vitae Researrch Center LLC, Miami, Florida
  - University of Miami, Miami, Florida
  - Miami Jewish Health Systems, Inc., Miami, Florida
  - United Health Research Corp. #1, Miami, Florida
  - United Health Research Corp. #2, Miami, Florida
  - Advanced Medical Center Group, Miami, Florida
  - Future Care Solution, LLC, Miami, Florida
  - Reliant Medical Research LLC Site #811, Miami, Florida
  - Hope Research Network LLC Site #773, Miami, Florida
  - Clinical Research Associates of South Florida #1, Miami, Florida
  - Clinical Research Associates of South Florida #2, Miami, Florida
  - Coral Research Clinic Corp, Miami, Florida
  - P&S RESEARCH, LLC. Site #805, Miami, Florida
  - Pharmax Research of South Florida, Miami, Florida
  - Kendall Research Institute, Miami, Florida
  - Nuovida Research Center Corp., Miami, Florida
  - New Med Research, Inc Site #812, Miami Gardens, Florida
  - Collier Neurologic Specialists, LLC, Naples, Florida
  - Naples Research, Inc, Naples, Florida
  - Bayside Clinical Research Site #556, New Port Richey, Florida
  - Research Centers of America, LLC, Oakland Park, Florida
  - Compass Research, LLC, Orlando, Florida
  - Combined Research Orlando Site #799, Orlando, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - IMIC Inc., Palmetto Bay, Florida
  - Innovation Medical Research Center Site #802, Palmetto Bay, Florida
  - University of West Florida, Pensacola, Florida
  - Neurostudies Inc. Site#796, Port Charlotte, Florida
  - Roskamp Institute, Sarasota, Florida
  - Olympian Clinical Research, Tampa, Florida
  - VICIS Clinical Research Inc. Site #777, Tampa, Florida
  - Compass Research North, LLC, The Villages, Florida
  - Neurology Research Institute Palm Beach, LLC #1, West Palm Beach, Florida
  - Neurology Research Institute Palm Beach, LLC #2, West Palm Beach, Florida
  - Florida Premier Research Institute, Winter Park, Florida
  - NeuroTrials Research Inc, Atlanta, Georgia
  - Columbus Research & Wellness Institute, INC, Columbus, Georgia
  - Medical Research & Health Education Foundation, Inc., Columbus, Georgia
  - NeuroStudies. Net, LLC, Decatur, Georgia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Josephson Wallack Munshower Neurology, PC, Indianapolis, Indiana
  - MidAmerica Neuroscience Research Foundation, Lenexa, Kansas
  - Four Rivers Clinical Research Inc., Paducah, Kentucky
  - The Samuel & Alexia Bratton Memory Clinic, Easton, Maryland
  - Mir Neurology, Hagerstown, Maryland
  - Alzheimer Disease Center Site #804, Braintree, Massachusetts
  - Boston Center for Memory, Newton, Massachusetts
  - Alzheimer's Disease Center, Quincy, Massachusetts
  - Onyx Clinical Research, LLC, Caro, Michigan
  - Michigan State University Department of Neurology, East Lansing, Michigan
  - Oakland Medical Research Site #762, Troy, Michigan
  - Galen Research, Chesterfield, Missouri
  - Millennium Psychiatric Associates, LLC, Creve Coeur, Missouri
  - The NeuroCognitive Institute, Mount Arlington, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - Dent Neurologic Institute, Amherst, New York
  - Integrative Clinical Trials LLC #1, Brooklyn, New York
  - Integrative Clinical Trials LLC #2, Brooklyn, New York
  - Columbia University Medical Center, New York, New York
  - Manhattan Behavioral Medicine, PLLC, New York, New York
  - Eastside Comprehensive Medical Center, LLC, New York, New York
  - Nathan S. Kline Institute for Psychiatric Research #1, Orangeburg, New York
  - Nathan S. Kline Institute for Psychiatric Research #571, Orangeburg, New York
  - University of Rochester Medical Center, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Burke Rehabilitation Hospital, White Plains, New York
  - Herbert Harris, Md, Phd, Pa, Chapel Hill, North Carolina
  - ANI Neurology PLLC dba Alzheimer's Memory Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Neurology and Neuroscience Associates, Inc., Akron, Ohio
  - Insight Clinical Trials, LLC Site #570, Beachwood, Ohio
  - Valley Medical Research Site #788, Centerville, Ohio
  - Valley Medical Research, Centerville, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - Cleveland Clinic Lou Ruvo Center for Brain Health at Lakewood Hospital, Lakewood, Ohio
  - NorthStar Medical Research Site #778, Middleburg Heights, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Oklahoma Clinical Research Center, Oklahoma City, Oklahoma
  - Heritage Valley Medical Group, Inc., Beaver, Pennsylvania
  - Abington Neurological Associates, LTD, Willow Grove, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - RH Johnson VA Medical Center, Charleston, South Carolina
  - Roper St. Francis Healthcare, Charleston, South Carolina
  - BG Neurology, Spartanburg, South Carolina
  - Texas Neurology, P.A., Dallas, Texas
  - Neurology Consultants of Dallas, PA, Dallas, Texas
  - University Texas Southwestern Medical Center, Dallas, Texas
  - InSite Clinical Research Site #576, DeSoto, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Neurological Institute, Houston, Texas
  - PRX Research Site #825, Mesquite, Texas
  - Texas Medical Research Associates, L.L.C., San Antonio, Texas
  - Ericksen Research and Development, Clinton, Utah
  - Pharmaceuticals Research Associates, Inc., Salt Lake City, Utah
  - Clinical Neuroscience Research Associates, Inc. dba The Memory Clinic, Bennington, Vermont
  - Neuropsychiatric Associates, Woodstock, Vermont
  - Veteran Affairs Medical Center, Salem Virginia, Salem, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Core Clinical Research Site #772, Everett, Washington
  - IPC Research, Waukesha, Wisconsin
- Bulgaria (7):
  - Center for Mental Health - Ruse, Rousse
  - Mental Health Centre Prof. Nikola Shipkovenski Site #713, Sofia
  - Medical Center Sveti Naum Site #707, Sofia
  - Vrach and Sv. Sv. Kuzma and Damian Site #710, Sofia
  - University Multiprofile Hospital for Active Treatment Alexandrovska Site #704, Sofia
  - Medical Center Mladost-M, Varna
  - Medica Plus Medical Center, Veliko Tarnovo
- Dr. Alexander McIntyre Inc., Penticton, Canada
- Czechia (11):
  - Fakultni Nemocnice u sv. Anny v Brne Site #722, Brno
  - Fakultní Nemocnice Hradec Králové Site #724, Hradec Kralové
  - NeuropsychiatrieHK Site #729, Hradec Kralové
  - Brain-Soultherapy, Kladno
  - Námestí národního odboje 692 Site #723, Kutná Hora
  - A-Shine s.r.o. Site #731, Pilsen
  - AD71, Prague
  - Clintrial, Prague
  - Neurologicka Ambulance - Forbeli, Prague
  - Neuropsychiatrie Site #726, Prague
  - Vestra Clinics, Rychnov nad Kněžnou
- France (3):
  - Centre Hospitalier Universitaire de Saint-Étienne - Hôpital Nord Site #535, Saint-Etienne, Auvergne-Rhône-Alpes
  - Centre Hospitalier Universitaire Dijon Bourgogn Site #536, Dijon
  - Centre Hospitalier Universitaire Toulouse - Casselardit Ancely Site #533, Toulouse
- Hungary (6):
  - Dr. Kenessey Albert Kórház-Rendelőintézet, Balassagyarmat
  - Pszichiatriai es Pszichiatriai Rehabilitacios Osztaly Site #586, Budapest
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Kenezy Gyula Egyetemi Korhaz, Debrecen
  - Dr. Mathe es Tarsa Beteti Tarsasag Site #593, Kalocsa
  - PsychoTech Clinical Research Site# 580, Pécs
- Italy (3):
  - Azienda Ospedaliera Sant'Andrea Site #606, Roma
  - Fondazione Policlinico Tor Vergata Site #609, Roma
  - Fondazione Santa Lucia - Istituto di Ricovero e Cura a Carattere Scientifico, Roma
- Poland (12):
  - Twoja Przychodnia - Centrum Medyczne Nowa Sol Site #757, Nowa Sól, Lubusz Voivodeship
  - RCMed Oddział Sochaczew Site #510, Sochaczew, Masovian Voivodeship
  - Ksiedza Hugona Kollataja 9, Bydgoszcz
  - Care Clinic Clinical Research Site #750, Katowice
  - Wielospecjalistyczna Poradnia Lekarska Synapsis Site #741, Katowice
  - Krakowska Akademia Neurologii Site #740, Krakow
  - Malopolskie Centrum Medyczne Site #747, Krakow
  - Medycyna Milorzab Site #743, Lodz
  - Solumed Centrum Medyczne Site #753, Poznan
  - Centrum Medyczne Euromedis, Szczecin
  - Centrum Medyczne NeuroProtect Site #742, Warsaw
  - ClinHouse Centrum Medyczne, Zabrze
- South Africa (5):
  - ACF Neurological Services, Cape Town
  - Cape Trial Centre, Cape Town
  - Flexivest Fourteen Research Centre, Cape Town
  - Apollo Clinical Research Site #623, Johannesburg
  - Medical and Dental Centre, Rosebank
- Spain (8):
  - Accellacare Alcobendas, Alcobendas
  - Fundació ACE, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Macarena Site #649, Seville
  - Complejo Asistencial de Zamora Hospital Virgen de la Concha, Zamora
  - Hospital Viamed Montecanal Site #643, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects took part in the study at 217 clinical sites in the North America and Europe from 13 November 2015 to 06 September 2024.
Pre-assignment Details: Of the 1197 subjects who were enrolled for the study, 1191 subjects received the study treatment, and 6 subjects did not receive the study drug. All eligible subjects received AVP-786-42.63/4.9, AVP-786-28/4.9, or AVP-786-18/4.9 depending on the last treatment received in the preceding study 15-AVP-786-301, 15-AVP-786-302, and 17-AVP-786-305.
Groups:
- AVP-786 18 18 Milligrams (mg): Participants who received AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) capsules in the previous studies 15-AVP-786-301 (NCT02442765), 15-AVP-786-302 (NCT02442778), or 17-AVP-786-305 (NCT03393520) continued to receive AVP-786-18 (d6-DM 18 mg/Q 4.9 mg), capsules, twice a day for 52 weeks in the current study.
Period: Overall Study
Arm/Group | AVP-786 18 18 Milligrams (mg) | AVP-786 28 mg | AVP-786 42.63 mg
Started | 166 | 517 | 514
Completed | 109 | 332 | 324
Not Completed | 57 | 185 | 190
Not completed — Adverse Event | 10 | 27 | 27
Not completed — Death | 2 | 13 | 10
Not completed — Lack of Efficacy | 1 | 10 | 6
Not completed — Lost to Follow-up | 2 | 4 | 5
Not completed — Non-compliance With Study Drug | 2 | 2 | 3
Not completed — Physician Decision | 1 | 8 | 13
Not completed — Protocol Deviation | 0 | 0 | 1
Not completed — Study Subject Withdrawal by Parent or Guardian | 14 | 36 | 22
Not completed — Study Terminated by Sponsor | 4 | 35 | 58
Not completed — Trial Site Terminated by Sponsor | 6 | 4 | 5
Not completed — Withdrawal by Subject | 11 | 29 | 25
Not completed — Reason not Specified | 4 | 16 | 10
Not completed — Enrolled Participants Who Did Not Receive Study Medications | 0 | 1 | 5

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received the study treatment.
Groups:
- AVP-786 18 mg: Participants who received AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) capsules in the previous studies 15-AVP-786-301 (NCT02442765), 15-AVP-786-302 (NCT02442778), or 17-AVP-786-305 (NCT03393520) continued to receive AVP-786-18 (d6-DM 18 mg/Q 4.9 mg), capsules, twice a day for 52 weeks in the current study.
- Total: Total of all reporting groups
Arm/Group | AVP-786 18 mg | AVP-786 28 mg | AVP-786 42.63 mg | Total
Number analyzed (Participants) | 166 | 516 | 509 | 1191
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.1 (8.1) | 75.6 (7.9) | 75.0 (7.5) | 75.1 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 286 | 295 | 676
  Male | 71 | 230 | 214 | 515
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 151 | 473 | 476 | 1100
  Race: Black or African American | 13 | 29 | 24 | 66
  Race: Asian | 2 | 4 | 2 | 8
  Race: American Indian or Alaska Native | 0 | 1 | 0 | 1
  Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Race: Other | 0 | 4 | 2 | 6
  Race: Missing | 0 | 4 | 5 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 69 | 215 | 278 | 562
  Ethnicity: Not Hispanic or Latino | 97 | 297 | 226 | 620
  Ethnicity: Missing | 0 | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE)is any untoward medical occurrence or unintended change (e.g. physical, psychological, or behavioral), including inter-current illness, whether considered related to treatment or not. An AE can therefore be any unfavorable and unintended sign (including any clinically significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A TEAE is defined as an AE that occurred or worsened after the first dose of study treatment up until 30 days after last dose.
Time Frame: From first dose of study drug (in current study) up to 3 months after last dose of study drug (up to Week 64)
Population: Safety population included all participants who received the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | AVP-786 18 mg | AVP-786 28 mg | AVP-786 42.63 mg
Number analyzed (Participants) | 166 | 516 | 509
Participants | 109 | 304 | 292

2. Primary Outcome: Number of Participants With Serious TEAE
Description: A serious adverse event (SAE) is any AE occurring at any dose that results in death, life-threatening experience, persistent or significant disability/incapacity, in-patient hospitalization or prolongation of hospitalization or congenital anomaly/birth defect. A serious TEAE is defined as AE that occurred or worsened after the first dose of study treatment up until 30 days after last dose.
Time Frame: From first dose of study drug (in current study) up to 3 months after last dose of study drug (up to Week 64)
Population: Safety population included all participants who received the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | AVP-786 18 mg | AVP-786 28 mg | AVP-786 42.63 mg
Number analyzed (Participants) | 166 | 516 | 509
Participants | 22 | 75 | 70

3. Primary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Test Abnormalities
Description: Laboratory assessments included clinical chemistry (alanine aminotransferase, albumin, alkaline phosphatase, aspartate aminotransferase, bilirubin, blood urea nitrogen, calcium, carbon dioxide, cholesterol, creatinine kinase, creatinine, gamma glutamyl transferase, glucose, lactate dehydrogenase, magnesium, protein, potassium, sodium, triglycerides and uric acid), hematology (basophils, eosinophils/leukocytes, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, lymphocytes/leukocytes, monocytes, monocytes/leukocytes, neutrophils/leukocytes, platelets). Number of participants with clinically significant laboratory test abnormalities were reported as per criteria defined in statistical analysis plan (SAP). The categories with at least one participant with potentially clinically significant laboratory values are reported.
Time Frame: Baseline (current study) up to 52 weeks
Population: Safety population included all participants who received the study treatment. 'Overall number analyzed' indicates the unique participants who were evaluated for this outcome measure. 'Number analyzed' indicates the number of participants evaluable for the specific category.
Measure: Count of Participants; unit: Participants
Arm/Group | AVP-786 18 mg | AVP-786 28 mg | AVP-786 42.63 mg
Number analyzed (Participants) | 166 | 516 | 509
Participants
  Alanine Aminotransferase (units per litre {U/L}): ≥3X ULN: number analyzed (Participants) | 164 | 510 | 508
  Alanine Aminotransferase (units per litre {U/L}): ≥3X ULN | 1 | 0 | 1
  Albumin (grams per litre {g/L}): ≤26 g/L: number analyzed (Participants) | 164 | 510 | 508
  Albumin (grams per litre {g/L}): ≤26 g/L | 3 | 1 | 2
  Albumin (g/L): ≥60 g/L: number analyzed (Participants) | 164 | 510 | 508
  Albumin (g/L): ≥60 g/L | 1 | 0 | 0
  Alkaline Phosphatase (U/L): ≥3X ULN: number analyzed (Participants) | 164 | 510 | 508
  Alkaline Phosphatase (U/L): ≥3X ULN | 1 | 0 | 1
  Aspartate Aminotransferase (U/L): ≥3X ULN: number analyzed (Participants) | 164 | 510 | 507
  Aspartate Aminotransferase (U/L): ≥3X ULN | 2 | 0 | 0
  Bilirubin (micromoles per liter {umol/L}): ≥1.5X ULN: number analyzed (Participants) | 164 | 510 | 508
  Bilirubin (micromoles per liter {umol/L}): ≥1.5X ULN | 0 | 2 | 4
  Blood Urea Nitrogen (millimoles per liter {mmol/L}): ≥10.71 mmol/L: number analyzed (Participants) | 158 | 450 | 398
  Blood Urea Nitrogen (millimoles per liter {mmol/L}): ≥10.71 mmol/L | 19 | 78 | 63
  Calcium (mmol/L): ≤1.75 mmol/L: number analyzed (Participants) | 164 | 508 | 508
  Calcium (mmol/L): ≤1.75 mmol/L | 0 | 1 | 0
  Calcium (mmol/L): ≥3.0 mmol/L: number analyzed (Participants) | 164 | 508 | 508
  Calcium (mmol/L): ≥3.0 mmol/L | 0 | 1 | 0
  Carbon Dioxide (mmol/L): >40 mmol/L: number analyzed (Participants) | 164 | 510 | 508
  Carbon Dioxide (mmol/L): >40 mmol/L | 0 | 0 | 1
  Cholesterol (mmol/L): ≥7.77 mmol/L: number analyzed (Participants) | 164 | 509 | 508
  Cholesterol (mmol/L): ≥7.77 mmol/L | 7 | 19 | 18
  Creatine Kinase (U/L): ≥3X ULN: number analyzed (Participants) | 164 | 507 | 505
  Creatine Kinase (U/L): ≥3X ULN | 2 | 4 | 4
  Creatinine (umol/L): >132.6 umol/L: number analyzed (Participants) | 164 | 510 | 508
  Creatinine (umol/L): >132.6 umol/L | 8 | 53 | 26
  Gamma Glutamyl Transferase (U/L): ≥60 U/L: number analyzed (Participants) | 164 | 501 | 488
  Gamma Glutamyl Transferase (U/L): ≥60 U/L | 13 | 52 | 51
  Glucose (mmol/L): ≤2.775 mmol/L: number analyzed (Participants) | 164 | 510 | 508
  Glucose (mmol/L): ≤2.775 mmol/L | 3 | 9 | 4
  Glucose (mmol/L): ≥11.1 mmol/L: number analyzed (Participants) | 164 | 510 | 508
  Glucose (mmol/L): ≥11.1 mmol/L | 22 | 71 | 79
  Lactate Dehydrogenase (U/L): ≥3X ULN: number analyzed (Participants) | 164 | 507 | 505
  Lactate Dehydrogenase (U/L): ≥3X ULN | 0 | 1 | 2
  Magnesium (mmol/L): <0.37 mmol/L: number analyzed (Participants) | 164 | 505 | 503
  Magnesium (mmol/L): <0.37 mmol/L | 1 | 1 | 0
  Magnesium (mmol/L): >1.23 mmol/L: number analyzed (Participants) | 164 | 505 | 503
  Magnesium (mmol/L): >1.23 mmol/L | 0 | 0 | 1
  Potassium (mmol/L): ≤3.0 mmol/L: number analyzed (Participants) | 164 | 510 | 507
  Potassium (mmol/L): ≤3.0 mmol/L | 2 | 4 | 2
  Potassium (mmol/L): ≥5.5 mmol/L: number analyzed (Participants) | 164 | 510 | 507
  Potassium (mmol/L): ≥5.5 mmol/L | 6 | 32 | 34
  Protein (g/L): ≤50 g/L: number analyzed (Participants) | 164 | 510 | 508
  Protein (g/L): ≤50 g/L | 3 | 0 | 4
  Sodium (mmol/L): ≤130 mmol/L: number analyzed (Participants) | 164 | 510 | 508
  Sodium (mmol/L): ≤130 mmol/L | 6 | 13 | 12
  Sodium (mmol/L): ≥155 mmol/L: number analyzed (Participants) | 164 | 510 | 508
  Sodium (mmol/L): ≥155 mmol/L | 0 | 1 | 2
  Triglycerides (mmol/L): >3.39 mmol/L: number analyzed (Participants) | 164 | 508 | 508
  Triglycerides (mmol/L): >3.39 mmol/L | 25 | 61 | 73
  Uric Acid (umol/L) (Female): ≥505.58 umol/L: number analyzed (Participants) | 94 | 282 | 295
  Uric Acid (umol/L) (Female): ≥505.58 umol/L | 3 | 22 | 14
  Uric Acid (umol/L) (Male): ≥624.54 umol/L: number analyzed (Participants) | 70 | 226 | 213
  Uric Acid (umol/L) (Male): ≥624.54 umol/L | 0 | 3 | 3
  Basophils (10^9/L): >0.3 x10^9/L: number analyzed (Participants) | 164 | 510 | 507
  Basophils (10^9/L): >0.3 x10^9/L | 0 | 1 | 1
  Eosinophils/Leukocytes (%): ≥10 %: number analyzed (Participants) | 164 | 509 | 505
  Eosinophils/Leukocytes (%): ≥10 % | 12 | 23 | 33
  Erythrocytes (10^12/L): ≤2.5 x10^12/L: number analyzed (Participants) | 164 | 510 | 507
  Erythrocytes (10^12/L): ≤2.5 x10^12/L | 0 | 0 | 1
  Erythrocytes (10^12/L): ≥7.0 x10^12/L: number analyzed (Participants) | 164 | 510 | 507
  Erythrocytes (10^12/L): ≥7.0 x10^12/L | 0 | 1 | 0
  Hematocrit (%): <0.3 proportion of 1.0: number analyzed (Participants) | 164 | 510 | 507
  Hematocrit (%): <0.3 proportion of 1.0 | 4 | 7 | 9
  Hematocrit (%): >0.5 proportion of 1.0: number analyzed (Participants) | 164 | 510 | 507
  Hematocrit (%): >0.5 proportion of 1.0 | 11 | 31 | 44
  Hemoglobin (g/L): <100 g/L: number analyzed (Participants) | 164 | 510 | 507
  Hemoglobin (g/L): <100 g/L | 5 | 15 | 15
  Hemoglobin (g/L): >180 g/L: number analyzed (Participants) | 164 | 510 | 507
  Hemoglobin (g/L): >180 g/L | 0 | 1 | 3
  Leukocytes (10^9/L): ≤2.8 x10^9/L: number analyzed (Participants) | 164 | 510 | 507
  Leukocytes (10^9/L): ≤2.8 x10^9/L | 2 | 7 | 3
  Leukocytes (10^9/L):≥16 x10^9/L: number analyzed (Participants) | 164 | 510 | 507
  Leukocytes (10^9/L):≥16 x10^9/L | 2 | 4 | 5
  Lymphocytes (10^9/L): ≤0.5 x10^9/L: number analyzed (Participants) | 164 | 510 | 507
  Lymphocytes (10^9/L): ≤0.5 x10^9/L | 0 | 4 | 7
  Lymphocytes (10^9/L): >4 x10^9/L: number analyzed (Participants) | 164 | 510 | 507
  Lymphocytes (10^9/L): >4 x10^9/L | 1 | 8 | 6
  Lymphocytes/Leukocytes (%): ≤10 %: number analyzed (Participants) | 164 | 509 | 505
  Lymphocytes/Leukocytes (%): ≤10 % | 6 | 30 | 21
  Lymphocytes/Leukocytes (%): ≥60 %: number analyzed (Participants) | 164 | 509 | 505
  Lymphocytes/Leukocytes (%): ≥60 % | 0 | 4 | 6
  Monocytes (10^9/L): >1 x10^9/L: number analyzed (Participants) | 164 | 510 | 507
  Monocytes (10^9/L): >1 x10^9/L | 7 | 27 | 23
  Monocytes/Leukocytes (%): ≥15 %: number analyzed (Participants) | 164 | 509 | 505
  Monocytes/Leukocytes (%): ≥15 % | 5 | 24 | 23
  Neutrophils/Leukocytes (%): ≤15 %: number analyzed (Participants) | 164 | 509 | 505
  Neutrophils/Leukocytes (%): ≤15 % | 0 | 1 | 1
  Platelets (10^9/L): ≤100 x10^9/L: number analyzed (Participants) | 164 | 510 | 507
  Platelets (10^9/L): ≤100 x10^9/L | 2 | 4 | 6
  Platelets (10^9/L): ≥700 x10^9/L: number analyzed (Participants) | 164 | 510 | 507
  Platelets (10^9/L): ≥700 x10^9/L | 0 | 0 | 1

4. Primary Outcome: Number of Participants With Potentially Clinically Significant 12-lead Electrocardiogram (ECG) Abnormalities
Description: A resting 12-lead ECG was performed for all the participants. ECG data included PR interval (milliseconds {msec}) and QTcF (msec) along with change from baseline in QTcF. Number of participants with potentially clinically significant ECG abnormalities was reported as per the criteria defined in SAP.
Time Frame: Baseline (current study) up to 52 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | AVP-786 18 mg | AVP-786 28 mg | AVP-786 42.63 mg
Number analyzed (Participants) | 166 | 516 | 509
Participants
  PR Interval Value (males and females): >200 to ≤220 msec: number analyzed (Participants) | 162 | 503 | 492
  PR Interval Value (males and females): >200 to ≤220 msec | 21 | 66 | 60
  PR Interval Value (males and females): >220 to ≤250 msec: number analyzed (Participants) | 162 | 503 | 492
  PR Interval Value (males and females): >220 to ≤250 msec | 13 | 33 | 28
  PR Interval Value (males and females): >250 msec: number analyzed (Participants) | 162 | 503 | 492
  PR Interval Value (males and females): >250 msec | 5 | 13 | 9
  QTcF Value (males): >450 to ≤480 msec: number analyzed (Participants) | 68 | 222 | 207
  QTcF Value (males): >450 to ≤480 msec | 9 | 28 | 23
  QTcF Value (males): >480 to ≤500 msec: number analyzed (Participants) | 68 | 222 | 207
  QTcF Value (males): >480 to ≤500 msec | 2 | 2 | 1
  QTcF Value (females): >470 to ≤485 msec: number analyzed (Participants) | 94 | 282 | 292
  QTcF Value (females): >470 to ≤485 msec | 3 | 12 | 10
  QTcF Value (females): >485 to ≤500 msec: number analyzed (Participants) | 94 | 282 | 292
  QTcF Value (females): >485 to ≤500 msec | 0 | 4 | 2
  QTcF Value (females): >500 msec: number analyzed (Participants) | 94 | 282 | 292
  QTcF Value (females): >500 msec | 0 | 1 | 1
  QTcF Change from Baseline (male and females): ≥30 msec: number analyzed (Participants) | 162 | 504 | 499
  QTcF Change from Baseline (male and females): ≥30 msec | 18 | 64 | 66
  QTcF Change from Baseline (male and females): ≥60 msec: number analyzed (Participants) | 162 | 504 | 499
  QTcF Change from Baseline (male and females): ≥60 msec | 1 | 5 | 5

5. Primary Outcome: Number of Participants With Any Abnormal, Clinically Significant Physical and Neurological Examination Finding
Description: The physical examination included assessments of head, eyes, ears, nose, throat, lymph nodes, skin, extremities, respiratory, gastrointestinal, musculoskeletal, cardiovascular, and nervous systems. The neurological examination included assessments of mental status, cranial nerves, motor system, reflexes, coordination, gait and station, and sensory system.
Time Frame: Baseline (current study), Week 52
Population: Safety population included all participants who received the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | AVP-786 18 mg | AVP-786 28 mg | AVP-786 42.63 mg
Number analyzed (Participants) | 166 | 516 | 509
Participants | 2 | 4 | 4

6. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities in Vital Signs
Description: Vital signs measurements included systolic blood pressure (SBP), diastolic blood pressure (DBP), and heart rate (HR). Blood pressure (i.e., SBP, DBP) and heart rate were measured in the supine and standing positions after the participant had been in each position for at least 5 and 3 minutes, respectively. Number of participants with clinically significant vital sign abnormalities were reported as per criteria defined in SAP. The categories with at least one participant with clinically significant vital signs abnormalities are reported here.
Time Frame: Baseline (current study) up to 52 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | AVP-786 18 mg | AVP-786 28 mg | AVP-786 42.63 mg
Number analyzed (Participants) | 166 | 516 | 509
Participants
  SBP: ≤90 and ≥20 decrease from baseline: number analyzed (Participants) | 164 | 507 | 509
  SBP: ≤90 and ≥20 decrease from baseline | 5 | 18 | 14
  SBP: >180 and ≥20 increase from baseline: number analyzed (Participants) | 164 | 507 | 509
  SBP: >180 and ≥20 increase from baseline | 0 | 6 | 4
  DBP: ≤50 and ≥15 decrease from baseline: number analyzed (Participants) | 164 | 507 | 509
  DBP: ≤50 and ≥15 decrease from baseline | 4 | 8 | 8
  DBP: ≥105 and ≥15 increase from baseline: number analyzed (Participants) | 164 | 507 | 509
  DBP: ≥105 and ≥15 increase from baseline | 2 | 3 | 8
  HR: ≤50 and ≥15 decrease from baseline: number analyzed (Participants) | 164 | 507 | 509
  HR: ≤50 and ≥15 decrease from baseline | 0 | 7 | 7
  HR: ≥120 and ≥15 increase from baseline: number analyzed (Participants) | 164 | 507 | 509
  HR: ≥120 and ≥15 increase from baseline | 0 | 4 | 1
  SBP ≥10 and HR ≥5 increase from baseline: number analyzed (Participants) | 164 | 507 | 509
  SBP ≥10 and HR ≥5 increase from baseline | 53 | 147 | 155
  DBP ≥5 and HR ≥5 increase from baseline: number analyzed (Participants) | 164 | 507 | 509
  DBP ≥5 and HR ≥5 increase from baseline | 61 | 239 | 225

7. Primary Outcome: Change From Baseline in the Sheehan Suicidality Tracking Scale (S-STS) Total Score at Week 64
Description: The S-STS is a prospective scale that assesses treatment-emergent suicidal thoughts and behaviors. This is a 20-item scale where each item (except item 17) of the S-STS is scored on a 5-point Likert scale as: 0 = Not at all, 1 = A little, 2 = Moderate, 3 = Very, 4 = Extremely. The S-STS total score is calculated by the sum of items 1a (if present), items 2-11, highest score of item 12 or 16, highest score of item 14 or 15, item 17 and 20. The total score ranges from 0 to 156 (If response to S-STS item 17 =yes, a score of 100 was added to the S-STS total score). Higher scores indicate greater severity of suicidal ideation and/or behavior. A negative change from baseline reflects a reduction in suicidal thoughts or behaviors over time.
Time Frame: Baseline (current study), Week 64
Population: Safety population included all participants who received the study treatment. 'Overall number of participants analyzed' indicates the number of participants evaluable for the outcome measure at the specified time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AVP-786 18 mg | AVP-786 28 mg | AVP-786 42.63 mg
Number analyzed (Participants) | 92 | 276 | 304
score on a scale | -0.0 (0.1) | 0.0 (0.1) | -0.0 (0.1)

8. Primary Outcome: Change From Baseline in the Mini-Mental State Examination (MMSE) Score at Week 52
Description: The MMSE is a brief questionnaire that is used to assess cognitive impairment and severity of cognitive impairment. The MMSE scale comprises 11 questions or simple tasks concerning orientation, memory, attention, and language to evaluate a participant's cognitive state and are scored as follows: Orientation to Time - 0 to 5; Orientation to Place - 0 to 5; Registration - 0 to 3; Attention and Calculation - 0 to 5; Recall - 0 to 3; Naming - 0 to 2; Repetition - 0 to 1; Comprehension - 0 to 3; Reading - 0 to 1; Writing - 0 to 1; Drawing - 0 to 1. The total score was calculated by summing all of the item scores and ranges from 0 to 30. Higher scores indicate milder cognitive impairment. Negative change from baseline indicates decline in cognitive performance.
Time Frame: Baseline (current study), Week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AVP-786 18 mg | AVP-786 28 mg | AVP-786 42.63 mg
Number analyzed (Participants) | 121 | 372 | 366
score on a scale | -0.8 (4.6) | -0.7 (4.9) | -0.1 (4.1)

9. Primary Outcome: Change From Baseline in the Epworth Sleepiness Scale (ESS) Score at Week 52
Description: The ESS is an 8-item questionnaire that is used to measure sleepiness by rating the probability of falling asleep on 8 different situations that most people engage in during the day. The 8 questions are rated on a 4-point scale (0 to 3) where 0 = would never doze, 1 = slight chance of dozing, 2 = moderate chance of dozing, and 3 = high chance of dozing. The scores are summed to give an overall score of 0 to 24. A total score of 0 to 9 is considered to be normal. Higher score indicates greater daytime sleepiness. Negative change from baseline indicate improvement in daytime sleepiness.
Time Frame: Baseline (current study), Week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AVP-786 18 mg | AVP-786 28 mg | AVP-786 42.63 mg
Number analyzed (Participants) | 83 | 297 | 338
score on a scale | -0.01 (4.43) | 0.07 (4.39) | 0.50 (3.93)

10. Secondary Outcome: Change From Baseline in the Cohen-Mansfield Agitation Inventory (CMAI) Composite Score at Week 64
Description: The CMAI is used to assess the frequency of manifestations of agitated behaviors in elderly persons. It consists of 29 agitated behaviors that are further categorized into distinct agitation syndromes, also known as CMAI factors of agitation. These distinct agitation syndromes include aggressive behavior, physically nonaggressive behavior, and verbally agitated behavior. Each of the 29 items is rated on a 7-point scale of frequency (1 = never, 2 = less than once a week but still occurring, 3 = once or twice a week, 4 = several times a week, 5 = once or twice a day, 6 = several times a day, 7 = several times an hour). The ratings are based on the 2 weeks preceding assessment of the CMAI. Higher scores indicate higher frequency of agitated behaviours while lower scores indicate lower frequency of agitated behaviours.
Time Frame: Baseline (current study), Week 64
Population: Due to discontinuation of development of the AVP-786 compound, no data was collected and analyzed as planned for this pre-specified secondary efficacy outcome measure as noted in the SAP. Only safety data was collected and analyzed.
Arm/Group | AVP-786 18 mg | AVP-786 28 mg | AVP-786 42.63 mg
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Change From Baseline in the Agitation/Aggression, Irritability/Lability, and Aberrant Motor Behavior Domain Scores of the Neuropsychiatric Inventory (NPI) at Week 52
Description: The NPI is a validated clinical instrument used to assess neuropsychiatric symptoms. It evaluates 12 neuropsychiatric symptom domains including delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, aberrant motor behavior, sleep and nighttime behavioral disorders, and appetite/eating disorders. Each symptom domain is rated by the caregiver based on the frequency (1 to 4) and severity (1 to 3) of symptoms, and a composite domain score is calculated by multiplying frequency and severity (range: 1-12). Additionally, caregiver distress for each positive symptom domain is rated on a 6-point scale (0 = not at all distressing, 5 = extremely distressing). In this study, the three NPI domains assessed were agitation/aggression, irritability/lability, and aberrant motor behavior. Higher scores indicate greater severity and frequency of neuropsychiatric symptoms.
Time Frame: Baseline (current study), Week 52
Population: as for outcome 10
Arm/Group | AVP-786 18 mg | AVP-786 28 mg | AVP-786 42.63 mg
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Change From Baseline in the Modified Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change-Agitation (mADCS-CGIC-Agitation) Score at Week 64
Description: The mADCS-CGIC-Agitation is used to assess agitation in individuals with Alzheimer's disease. It includes questions focused on agitation and uses a semi-structured interview format involving both the participant and their caregiver. The clinician rates the participant's overall clinical status using a 7-point scale: 1 = marked improvement, 2 = moderate improvement, 3 = minimal improvement, 4 = no change, 5 = minimal worsening, 6 = moderate worsening, and 7 = marked worsening. Lower scores indicate improvement in agitation symptoms, while higher scores indicate worsening.
Time Frame: Baseline (current study), Week 64
Population: as for outcome 10
Arm/Group | AVP-786 18 mg | AVP-786 28 mg | AVP-786 42.63 mg
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Change From Baseline in the Clinical Global Impression of Severity of Illness (CGIS)-Agitation Domain Score at Week 52
Description: The CGIS is an observer-rated scale that measures illness severity. The CGIS-Agitation is a 7-point (1-7) scale (1 = normal, not at all ill; 7 = extremely ill) that assessed the severity of agitation in this study. Higher scores indicate severe agitation, while the lower scores indicate little or no agitation.
Time Frame: Baseline (current study), Week 52
Population: as for outcome 10
Arm/Group | AVP-786 18 mg | AVP-786 28 mg | AVP-786 42.63 mg
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Change From Baseline in the Patient Global Impression of Change (PGIC) Score at Week 52
Description: The PGIC is a 7-point scale used to assess perceived treatment response, as evaluated by the participant's caregiver. The caregiver rates the overall change in the participant's condition since the start of treatment. The PGIC score ranges from 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. Lower scores reflect greater improvement, while higher scores indicate worsening of the participant's condition.
Time Frame: Baseline (current study), Week 52
Population: as for outcome 10
Arm/Group | AVP-786 18 mg | AVP-786 28 mg | AVP-786 42.63 mg
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Change From Baseline in the Dementia Quality of Life (DEMQOL) Score at Week 52
Description: The DEMQOL is a validated scale used to assess health-related quality of life in individuals with dementia and their caregivers. It includes two versions: a 28-item version completed by the participant (DEMQOL), and a 31-item proxy version completed by the caregiver (DEMQOL-proxy). Each item is rated using a 4-point scale to reflect the frequency or severity of health-related concerns: 1 = A lot, 2 = Quite a bit, 3 = A little, 4 = Not at all. Total score is derived by sum of all item scores, excluding item 29 of DEMQOL and item 32 of DEMQOL-proxy. Lower scores indicate better quality of life.
Time Frame: Baseline (current study), Week 52
Population: as for outcome 10
Arm/Group | AVP-786 18 mg | AVP-786 28 mg | AVP-786 42.63 mg
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Change From Baseline in the Resource Utilization in Dementia (RUD) Score at Week 52
Description: The RUD is a standardized tool used to estimate healthcare costs associated with dementia. It assesses the use of both formal and informal (e.g., hospitalizations, doctor visits, living assistance, and unprofessional caregiver time) healthcare resources. The instrument is administered as a semi-structured interview with the participant's primary caregiver. It consists of two main sections: one evaluates the caregiver's burden, including lost work and leisure time, and the other documents the participant's use of healthcare services. Total healthcare costs are calculated by multiplying the quantity of resources used (e.g., number of doctor visits, hours of caregiver, nights in accommodation) by unit costs. Higher estimated totals reflect greater economic impact associated with dementia care.
Time Frame: Baseline (current study), Week 52
Population: as for outcome 10
Arm/Group | AVP-786 18 mg | AVP-786 28 mg | AVP-786 42.63 mg
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Change From Baseline in the EuroQol 5-Dimension 5-Level (EQ-5D-5L) for Participants From Study 17-AVP-786-305 at Week 52
Description: The EQ-5D-5L is a standardized questionnaire used to assess health-related quality of life. It consists of two components: a descriptive system and the EuroQol Visual Analogue Scale (EQ VAS). The descriptive system covers five health dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on a 5-level scale: 1 = No problems, 2 = Slight problems, 3 = Moderate problems, 4 = Severe problems, 5 = Extreme problems. The EQ VAS component allows participants or caregivers to rate the individual's overall health on a vertical scale from 0 (the worst imaginable health state) to 100 (the best imaginable health state). Only participants from Study 17-AVP-786-305 with a MMSE score of 10 or higher at the baseline visit were planned to complete the participant-rated version.
Time Frame: Baseline (current study), Week 52
Population: as for outcome 10
Arm/Group | AVP-786 18 mg | AVP-786 28 mg | AVP-786 42.63 mg
Number analyzed (Participants) | 0 | 0 | 0

18. Other Pre Specified Outcome: Number of Participants Using Concomitant Medications
Description: Concomitant medications were defined as any medications taken on or after the date of first dose of study drug in Study 15-AVP-786-303 or that are ongoing concomitant medications from Studies 15-AVP-786-301, 15-AVP-786-302, 17-AVP-786-305, and 12-AVR-131.
Time Frame: Baseline (current study) up to 64 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From first dose of study drug (in current study) up to 3 months after last dose of study drug (up to Week 64)
Description: Safety population included all subjects who received the study treatment.
Arm/Group | AVP-786 18 mg | AVP-786 28 mg | AVP-786 42.63 mg
All-Cause Mortality (participants affected / at risk) | 4/166 | 22/516 | 16/509
Serious Adverse Events (participants affected / at risk) | 22/166 | 75/516 | 70/509
Other Adverse Events (participants affected / at risk) | 54/166 | 150/516 | 149/509
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AVP-786 18 mg (N=166) | AVP-786 28 mg (N=516) | AVP-786 42.63 mg (N=509)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 1
Bradycardia (Cardiac disorders) | 0 | 2 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 2
Cardiac arrest (Cardiac disorders) | 0 | 1 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 2
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 1 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 0 | 1
Pulmonary valve stenosis (Cardiac disorders) | 0 | 1 | 0
Keratitis (Eye disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 2
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Volvulus of small bowel (Gastrointestinal disorders) | 0 | 0 | 1
Death (General disorders) | 0 | 2 | 1
Asthenia (General disorders) | 0 | 0 | 1
Disease progression (General disorders) | 0 | 1 | 0
Inflammation (General disorders) | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 5 | 7
Pneumonia (Infections and infestations) | 1 | 3 | 8
COVID-19 (Infections and infestations) | 0 | 2 | 1
Cystitis (Infections and infestations) | 1 | 0 | 2
Pneumonia aspiration (Infections and infestations) | 1 | 2 | 0
Sepsis (Infections and infestations) | 2 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 0
Colonic abscess (Infections and infestations) | 0 | 0 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 1
Psoas abscess (Infections and infestations) | 0 | 0 | 1
Pyuria (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 12 | 5
Femur fracture (Injury, poisoning and procedural complications) | 0 | 3 | 3
Hip fracture (Injury, poisoning and procedural complications) | 0 | 4 | 2
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1
Intentional medical device removal by patient (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 1 | 0
Blood osmolarity increased (Investigations) | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0
QRS axis abnormal (Investigations) | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 5 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Syncope (Nervous system disorders) | 3 | 4 | 4
Dementia Alzheimer's type (Nervous system disorders) | 1 | 3 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 2
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 1
Unresponsive to stimuli (Nervous system disorders) | 0 | 1 | 1
Balance disorder (Nervous system disorders) | 0 | 1 | 0
Basal ganglia haematoma (Nervous system disorders) | 0 | 0 | 1
Brain hypoxia (Nervous system disorders) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
Dementia (Nervous system disorders) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1
Dysstasia (Nervous system disorders) | 1 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Neurodegenerative disorder (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 4 | 6 | 4
Mental status changes (Psychiatric disorders) | 0 | 0 | 4
Aggression (Psychiatric disorders) | 1 | 1 | 1
Delirium (Psychiatric disorders) | 0 | 2 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 2 | 0
Confusional state (Psychiatric disorders) | 0 | 2 | 0
Disturbance in social behaviour (Psychiatric disorders) | 0 | 1 | 0
Dysphemia (Psychiatric disorders) | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 2 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 4
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1
Neurogenic bladder (Renal and urinary disorders) | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 2
Orthostatic hypotension (Vascular disorders) | 1 | 1 | 0
Femoral artery aneurysm (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Peripheral artery aneurysm (Vascular disorders) | 0 | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 1 | 0
Peripheral embolism (Vascular disorders) | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AVP-786 18 mg (N=166) | AVP-786 28 mg (N=516) | AVP-786 42.63 mg (N=509)
Diarrhoea (Gastrointestinal disorders) | 10 | 28 | 26
Urinary tract infection (Infections and infestations) | 13 | 45 | 43
Contusion (Injury, poisoning and procedural complications) | 10 | 16 | 11
Fall (Injury, poisoning and procedural complications) | 27 | 79 | 60
Headache (Nervous system disorders) | 10 | 14 | 17
Agitation (Psychiatric disorders) | 10 | 32 | 39

LIMITATIONS AND CAVEATS:
The study was prematurely terminated due to discontinuation of development of the AVP-786 compound.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/32/NCT02446132/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/32/NCT02446132/SAP_001.pdf